CLINICAL TRIAL: NCT06941740
Title: Randomized Controlled Nutrition Trial on Reactive Hypoglycaemia on the Course of Memory and Attention Among Young Adults - Relevance of Chronotype
Brief Title: Effects of Reactive Hypoglycaemia on Cognition in Earlier or Later Chronotypes
Acronym: GlyCoBrainI2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anette Buyken (Other)
Collaborators: Paderborn University (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Anette Buyken, Prof. Dr., Paderborn University
Organization: Paderborn University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BU 1807/8-1-2
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: chronotype; breakfast; continuous glucose monitoring; MCTQ; memory; attention; cognition; body composition; glycaemic index; reactive hypoglycaemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: It is estimated that a maximum of 177 participants will need to be invited to obtain full data sets from 44 participants of an earlier chronotype and 44 of a later chronotype each completing the cross-over designed intervention study. The intervention study consists of the consumption of one of two low-GI beverages at 09:00 a.m., with one of these beverages ("glucose-fructose-sucrose beverage") inducing reactive hypoglycaemia and the other not ("isomaltulose beverage"). The participants will be randomly assigned to receive one of the two beverages on the first intervention day and the other on the second intervention day. The trial is a two-arm crossover study. Each participant serves as his or her own control, thus accounting for interindividual variations in diurnal glycaemic responses and cognitive performance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind, meaning that neither participants nor researchers know which of the two low-GI beverages they are consuming. Beverages will be pre-prepared by staff who are not involved in its provision.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-GI beverage causing reactive hypoglycaemia (Experimental): low-GI beverage causing reactive hypoglycaemia consisting of 75 g glucose-fructose-sucrose dissolved in 500 ml tap water
  Interventions: Other: immediate verbal memory after low glycemic index breakfast inducing no reactive hypoglycaemia; Other: immediate verbal memory after low glycemic index breakfast causing reactive hypoglycaemia
- low-GI beverage not inducing reactive hypoglycaemia (Experimental): low-GI beverage not inducing reactive hypoglycaemia consisting of 75 g isomaltulose dissolved in 500 ml tap water
  Interventions: Other: immediate verbal memory after low glycemic index breakfast inducing no reactive hypoglycaemia; Other: immediate verbal memory after low glycemic index breakfast causing reactive hypoglycaemia

INTERVENTIONS:
Other: immediate verbal memory after low glycemic index breakfast inducing no reactive hypoglycaemia — - Difference in immediate verbal memory after low GI breakfast without reactive hypoglycaemia at 90minutes
Other: immediate verbal memory after low glycemic index breakfast causing reactive hypoglycaemia — - Difference in immediate verbal memory after low GI breakfast causing reactive hypoglycaemia at 90 minutes

SUMMARY:
Studies suggest a link between lower postprandial glycaemic response and better cognitive performance in children, adolescents, and young adults, though evidence remains inconclusive. High glycaemic index (GI) meals quickly raise blood glucose, potentially causing reactive hypoglycaemia (glucose levels below baseline) and harming cognitive performance, especially in the late postprandial period, particularly after 120 minutes. Young adults may be more sensitive to these cognitive effects due to morning circadian misalignment, as their sleep midpoint (chronotype) is biologically most delayed. Recent research suggests that those with later chronotypes do not display the known circadian decline in glucose tolerance as indicated by equally high glycaemic responses to the same high GI meal in the morning or the evening. Eating breakfast "against the inner clock" may harm glycaemic response, particularly for those with a later chronotype. Those with morning circadian misalignment may also limit breakfast to beverages. Reactive hypoglycaemia commonly follows beverage consumption, especially soft drinks, energy drinks, glucose solutions, and low-GI fruit juices, occurring within 60 minutes after consumption. Later chronotypes may be more prone to reactive hypoglycaemia from drinks, harming cognition. This nutrition trial aims to investigate (I) the effects of breakfast-induced reactive hypoglycaemia on memory and attention in young, healthy, non-obese university students and (II) the relevance of chronotype to hypoglycaemia occurrence. To study reactive hypoglycaemia, a low GI beverage will be used, causing hypoglycaemia despite a low glycaemic response. Two samples will be examined: students of early and late chronotype. Postprandial insulin and cortisol changes will be analyzed, as improved insulin sensitivity and cortisol levels seem to affect cognition. From October 2024 to January 2025, 356 students (ages 18-25) enrolled in the GlyCoBrain Observational study (ID: NCT06679088) and were screened for chronotypes at Paderborn University. Participants with extreme chronotypes will be invited to this crossover study. Power calculations indicated a sample of 88 participants who complete both intervention days. They will consume a low-GI beverage at 9 a.m. causing reactive hypoglycaemia (glucose-fructose-sucrose solution) or a non-hypoglycaemia causing beverage (isomaltulose® solution) and undergo repeated cognitive assessments for the following 180 minutes.

DETAILED DESCRIPTION:
Studies in young adults indicate beneficial effects of a low-glycaemic index (GI) breakfast on cognitive performance. A meta-analysis of 17 studies revealed the benefits of a low-glycaemic (GL) load breakfast on immediate verbal memory only in the late postprandial period. No overall effect on attention in adults was reported, yet advantages for attention in children, adolescents, and young adults were suggested. Mechanisms explaining the time-dependent benefits of a low GL breakfast are not fully understood. The provision of glucose to the brain is currently discussed as a central mechanism linking meal GI/GL to cognition. Glucose is required for cognitive efforts as evidenced by decreases in local extracellular glucose concentrations in the activated brain area. Key neurotransmitter synthesis in the brain needs glucose. Glucose metabolism may influence memory through tryptophan utilization and serotonin concentrations. The memory-enhancing effect of glucose may require relatively constant blood glucose levels in the brain rather than high glucose amounts per se. Hence, whilst high GI foods elicit a transient increase in blood glucose levels, low-GI foods will result in a more sustained and longer-lasting provision of glucose. The late postprandial phase, when cognitive benefits of low GI/GL meals are most noticeable, coincides with the time after reactive hypoglycaemia following a high-GI meal. To disentangle the effects of dietary GI and reactive hypoglycaemia, it is prudent to examine beverages like fruit juices - characterized by a low GI, yet known to induce reactive hypoglycaemia even earlier postprandially. Accordingly, also detrimental effects on cognition should manifest earlier as observed for high-GI breakfast. Since recent work suggests that there may be an optimal blood glucose range for cognitive performance and that this optimal range may differ by cognitive domain, continuous glucose monitoring should be used in addition to the conventional measurement points directly before the cognitive test. However, benefits of low GI/GL breakfast for cognitive function have also been observed without differences in blood glucose levels. This may be attributable to an acutely improved postprandial insulin sensitivity and/or lower cortisol levels elicited by low-GI meals. Accordingly, concomitant examinations of all three factors, i.e. glucose, insulin and cortisol levels seem necessary to disentangle potential mechanisms. The above-mentioned meta-analysis also found greater benefits for individuals with better glucose tolerance, although age may confound this. Studies suggest that young adults with poorer glucose tolerance, even within the healthy range, may be more vulnerable to these effects. While glucose tolerance follows a circadian rhythm, being lowest in the evening due to reduced pancreatic β-cell function and insulin response, circadian misalignment-common among young adults with later chronotypes-can also impair glucose tolerance, even at breakfast, due to decreased insulin sensitivity. This misalignment, often caused by social jetlag, has been linked to obesity, type 2 diabetes, higher blood glucose, HbA1c levels, and an increased risk of depression. It remains unclear whether persons with later chronotypes are more susceptible to reactive hypoglycaemia after breakfast.

Hypothesis

1. Reactive hypoglycaemia in response to a low-GI beverage impairs memory and attention after approx. 90 minutes
2. Reactive hypoglycaemia after the consumption of low-GI beverage is more pronounced in healthy persons with a later chronotype
3. The adverse effect of a low-GI breakfast inducing reactive hypoglycaemia on memory and attention is particularly evident in those with later chronotype Aim This nutrition trial aims to investigate how low-GI beverages induce reactive hypoglycaemia and its effects on memory and attention after meals in postprandial phase. The investigators aim to explore the effects of chronotype in two student samples: those with earlier and later chronotypes. Further, the study investigate the relevance of chronotype for the postprandial course of glucose (including the occurrence of reactive hypoglycaemias), insulin and cortisol levels.

Methodology

Participants Healthy, German-speaking students at Paderborn University (early or late chronotype)

Sample size calculation:

Sample size calculation based on the difference in immediate memory and the study rated best in terms of quality in the meta-analysis. Given a standard deviation of 3.6 and 4.3 in both groups, and a standardized mean difference of 0.31 for people with a better glucose tolerance (corresponding to mean difference of 1.12) 44 participants are required in the smallest subgroup with a given power of 80% and alpha of 0.05 considering a correlation of 0.8 between both measurements (calculated with STATA, vers. 17.0). The investigator assume that 66% of invited students will participate and that 75% of those will complete the study. Hence, to have the full data set of 88 persons (44 with an early chronotype and 44 with a late chronotype) completing the trial, 117 need to start the trial and 177 people need to be invited from the GlyCoBrain Observational study which recruited 356 students from Paderborn University and screened for chronotype via MCTQ. Both chronotype samples have equal sex distribution.

Both samples will be invited to participate in the crossover nutrition trial, excluding smokers, shift workers or travelers of >2 time zones in the past 3 months, and persons taking methylphenidate or melatonin. Students will participate in 2 breakfast cognition tests, each after an overnight fast at 8 a.m. to be taken over 2 weeks including 1 week of wash-out. Participants will be assigned randomly to one of two sequence groups, differing only in the intervention sequence (isomaltulose® beverage, glucose-fructose-sucrose beverage or glucose-fructose-sucrose beverage, isomaltulose® beverage). Randomization lists are provided by an external statistical advisor from the University of Esbjerg stratified by sex and chronotype. A randomized list was generated for 4 groups, each with 30 slots, using a block randomization approach. The randomization was performed using STATA with 5 blocks, ensuring balance across the groups.

Participants will receive two different simple beverage breakfasts:

1. low-GI beverage causing reactive hypoglycaemia ("glucose-fructose-sucrose beverage") consisting of a 75 g glucose-fructose-sucrose mixture dissolved in 500 ml tap water
2. low-GI beverage inducing no reactive hypoglycaemia ("isomaltulose® beverage") consisting of 75 g isomaltulose dissolved in 500 ml tap water

The intervention follows a 2-week schedule:

Week 1: Participants are invited for preparation day 1 (Friday), during which a venous fasted blood sample is taken to determine fasting lipids, high-sensitivity-C-reactive protein, alanine aminotransferase and gamma-glutamyltransferase to metabolically characterize the recruited participants. To validate the previously determined chronotype in the GlyCoBrain Observational study, participants' chronotype will be assessed again using the Munich chronotype questionnaire. (MCTQ, © Roenneberg and co-workers, 2003). Body composition will be reassessed by Bioimpedance Analysis (mBCA 515, SECA, Germany) to estimate individual percentages of body fat, muscle mass, total body water and extracellular water. Body weight will be measured using the medical Body Composition Analyzer (mBCA). Body height will be measured using an ultrasound measuring station (seca 287 db). Waist circumference will be measured at the midpoint between the lower ribcage and hip bone of the exposed upper body.

Continuous glucose monitoring (CGM, G7, Dexcom, Inc., San Diego,CA) is activated, and an accelerometer will be used to measure movement and sleep/wake conditions (also allowing to corroborate chronotype). A standardized evening meal will be provided to be consumed in the evening before the intervention to avoid secondary meal effects e.g. caused by pulse consumption. Participants will be asked to perform a training session on the cognition battery (see below).

The actual intervention starts three to five days later at 8 a.m. with each day running as follows:

* Heart rate belt to measure the heart rate variability in combination with the fitness watch (Polar Electro, Finland).
* minimal invasive capillary blood samples collected at -40, 30, 80 and 140 minutes (in relation to the time point of drinking the beverage) will be used to determine glucose and insulin levels
* non-invasively cortisol samples from saliva at -40, 80 and 140 minutes
* continuous glucose measurements
* Cognition test at -30, 90 and 150 minutes
* test beverage breakfast including either glucose-fructose-sucrose or Isomaltulose to be drunk at time point 0, i.e. 09:00 a.m.
* other measurements: appetite, thirst and mood will be assessed at -40, 30, 80 and 140 minutes each using a validated visual analogue scale
* removal of all devices and provision of a voluntary breakfast at 180 minutes Glucose levels will be directly determined using HemoCue Glucose 201 RT Analyzer (HemoCue AB, Sweden). Plasma insulin concentration and cortisol concentration in saliva will be determined by an enzyme-linked immunosorbent assay using a kit from IBL/Tecan.

Week 2: Again, participants repeat the preparation day as before (day 2), except for BIA, MCTQ and venous blood sample measurements. The intervention then continues 3 to 5 days after the preparation day following the same time scale as on intervention day 1.

Cognition tests Assessment using the test battery is expected to last approximately 25 minutes in total each time. Tests will include a set of tests developed by the ALA Institute Bochum, that was applied in previous studies.

* (Delayed) verbal memory test (ability to correctly recall a total of 30 words immediately (recall) and after 20 minutes (delayed recall))
* Visual-spatial short-term working memory test (a Corsi-block tapping test equivalent, i.e., tapping a sequence of up to nine identical spatially separated blocks, sequentially increasing the difficulty by the number of presented blocks).
* Test of selective and sustained attention and visual scanning speed (a modified version of the d2 Test of attention, during which the reaction-specific signs within a series of presented signs will be assessed)
* Test of spatial attention and switching abilities between two different tasks (alternative version of the Trail Making Task)
* Test of tonic alertness (simple reaction time test)
* Test of inhibition, i.e. the ability to inhibit a prepotent response, using a flanker task. In each trial, three superposed triangles will be presented to the participants. The upper and lower triangles (flankers) will be pointing in the same direction but independent from the middle triangle (target). During the no-go trials, a circle replaces the target. The participants will be supposed to press the buttons left or right according to the direction of the target or not to react in the case of a no-go condition. Each trial will be categorized as compatible-go, incompatible-go or no-go.
* A dummy test to ensure that delayed recall starts exactly 20 minutes after the immediate recall

Statistical analysis Multilevel regression models will be employed to assess the effect of the interventions on immediate verbal memory at 90 minutes. Identical models will be used for the other cognitive outcomes. Interactions between the intervention effect and the chronotype will be tested, and stratified analyses based on the chronotype will be conducted. Further analyses will account for the sensitivity of insulin, and other factors such as cortisol, appetite, thirst and/or mood, to investigate whether the observed effects could be partially explained by these factors. Multilevel regression analyses with repeated measurements will assess the relevance of chronotype to reactive hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants of GlyCoBrain Observational Study
* Early or late chronotype (approx. lowest and highest quartile)

Exclusion Criteria:

* Students studying nutritional science or home economics (study programs of the study PI)
* Intermediate chronotypes
* Persons unwilling to abstain from smoking or cannabis use during the intervention period
* Persons unwilling to consume standard evening meals before intervention days
* BMI>30 kg/m² (diurnal variation in glycaemic control is known to be absent among persons with obesity) and <18.5 kg/m2 (since underweight is also known to affect glucose homeostasis)
* acute or permanent use of sleep-promoting medications (including herbal preparation):

  * medications: melatonin, diphenhydramine, doxylamine
  * herbal preparations: hops, St. John's wort, lemon balm, lavender, passionflower, Baldurat, Neurexan, cannabinoids
* Use of psychotropic medications (antidepressants, tranquillizers, antipsychotics)
* Use of methylphenidate (e.g. Ritalin, Medikinet, Concerta)
* Use of cannabinoids by prescription
* Continuous administration of antihistamines when discontinuation is not feasible during the intervention
* Use of herbal preparations affecting memory and concentration (e.g. ginkgo, ginseng, ashwagandha)
* Use of other medications (e.g. insulin, metformin, SGLT2 inhibitors, steroids, ACE inhibitors)
* Selected chronic diseases (depression and other mental disorders such as anxiety disorder, ADHD, diabetes mellitus (all types), prediabetes, blood clotting disorders (e.g., thrombocytopenia, haemophilia), eating disorders (e.g., anorexia, binge eating, bulimia), Chronic inflammatory bowel diseases, infectious diseases (HIV, hepatitis), Addiction disorders (e.g., alcohol, drug, or medication dependency)
* Pregnant and breastfeeding individuals
* Shift work or travel in the past 3 months across more than 2 time zones
* students with a pacemaker/defibrillator or cochlear implant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Difference in immediate memory between low-GI breakfast | On the first intervention day and after one week from -30 until 150 minutes after intervention focusing on 90 minutes (when reactive hypoglycaemia is expected to manifest)
  Computer-assisted cognition test

CONTACTS AND LOCATIONS:
Overall Officials: Lars Libuda, Prof. Dr., Prof. Dr., Principal Investigator — Paderborn University
Locations (1):
- Paderborn University, Paderborn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroder M, Muller K, Falkenstein M, Stehle P, Kersting M, Libuda L. Lunch at school and children's cognitive functioning in the early afternoon: results from the Cognition Intervention Study Dortmund Continued (CoCo). Br J Nutr. 2016 Oct;116(7):1298-1305. doi: 10.1017/S0007114516002932. Epub 2016 Sep 9. PMID 27608921
- [Background] Schroder M, Muller K, Falkenstein M, Stehle P, Kersting M, Libuda L. Short-term effects of lunch on children's executive cognitive functioning: The randomized crossover Cognition Intervention Study Dortmund PLUS (CogniDo PLUS). Physiol Behav. 2015 Dec 1;152(Pt A):307-14. doi: 10.1016/j.physbeh.2015.09.025. Epub 2015 Sep 30. PMID 26427889
- [Background] Stern RA, Arruda JE, Hooper CR, Wolfner GD, Morey CE. Visual analogue mood scales to measure internal mood state in neurologically impaired patients: Description and initial validity evidence. Aphasiology 1997;11(1):59-71.
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Deng Q, Haszard JJ, Conner TS, Rapsey C, Peng M, Venn BJ. Cognitive performance, mood and satiety following ingestion of beverages imparting different glycaemic responses: a randomised double-blind crossover trial. Eur J Clin Nutr. 2021 Apr;75(4):602-610. doi: 10.1038/s41430-020-00749-6. Epub 2020 Sep 17. PMID 32943769
- [Background] Lotti S, Pagliai G, Colombini B, Sofi F, Dinu M. Chronotype Differences in Energy Intake, Cardiometabolic Risk Parameters, Cancer, and Depression: A Systematic Review with Meta-Analysis of Observational Studies. Adv Nutr. 2022 Feb 1;13(1):269-281. doi: 10.1093/advances/nmab115. PMID 34549270
- [Background] Morris CJ, Yang JN, Garcia JI, Myers S, Bozzi I, Wang W, Buxton OM, Shea SA, Scheer FA. Endogenous circadian system and circadian misalignment impact glucose tolerance via separate mechanisms in humans. Proc Natl Acad Sci U S A. 2015 Apr 28;112(17):E2225-34. doi: 10.1073/pnas.1418955112. Epub 2015 Apr 13. PMID 25870289
- [Background] Saad A, Dalla Man C, Nandy DK, Levine JA, Bharucha AE, Rizza RA, Basu R, Carter RE, Cobelli C, Kudva YC, Basu A. Diurnal pattern to insulin secretion and insulin action in healthy individuals. Diabetes. 2012 Nov;61(11):2691-700. doi: 10.2337/db11-1478. Epub 2012 Jun 29. PMID 22751690
- [Background] Kennedy DO, Scholey AB. Glucose administration, heart rate and cognitive performance: effects of increasing mental effort. Psychopharmacology (Berl). 2000 Mar;149(1):63-71. doi: 10.1007/s002139900335. PMID 10789884
- [Background] Donohoe RT, Benton D. Cognitive functioning is susceptible to the level of blood glucose. Psychopharmacology (Berl). 1999 Aug;145(4):378-85. doi: 10.1007/s002130051071. PMID 10460314
- [Background] Lamport DJ, Chadwick HK, Dye L, Mansfield MW, Lawton CL. A low glycaemic load breakfast can attenuate cognitive impairments observed in middle aged obese females with impaired glucose tolerance. Nutr Metab Cardiovasc Dis. 2014 Oct;24(10):1128-36. doi: 10.1016/j.numecd.2014.04.015. Epub 2014 May 14. PMID 24925124
- [Background] Dye L, Gilsenan MB, Quadt F, Martens VE, Bot A, Lasikiewicz N, Camidge D, Croden F, Lawton C. Manipulation of glycemic response with isomaltulose in a milk-based drink does not affect cognitive performance in healthy adults. Mol Nutr Food Res. 2010 Apr;54(4):506-15. doi: 10.1002/mnfr.200900196. PMID 20140897
- [Background] Sanchez-Aguadero N, Recio-Rodriguez JI, Patino-Alonso MC, Mora-Simon S, Alonso-Dominguez R, Sanchez-Salgado B, Gomez-Marcos MA, Garcia-Ortiz L. Postprandial effects of breakfast glycaemic index on cognitive performance among young, healthy adults: A crossover clinical trial. Nutr Neurosci. 2020 Jan;23(1):1-7. doi: 10.1080/1028415X.2018.1461459. Epub 2018 Apr 12. PMID 29649949
- [Background] Nabb S, Benton D. The influence on cognition of the interaction between the macro-nutrient content of breakfast and glucose tolerance. Physiol Behav. 2006 Jan 30;87(1):16-23. doi: 10.1016/j.physbeh.2005.08.034. Epub 2005 Oct 12. PMID 16225896
- [Background] Benton D, Nabb S. Breakfasts that release glucose at different speeds interact with previous alcohol intake to influence cognition and mood before and after lunch. Behav Neurosci. 2004 Oct;118(5):936-43. doi: 10.1037/0735-7044.118.5.936. PMID 15506876
- [Background] Anderson JR, Maki KC, Palacios OM, Edirisinghe I, Burton-Freeman B, Spitznagel MB. Varying roles of glucoregulatory function measures in postprandial cognition following milk consumption. Eur J Nutr. 2021 Apr;60(3):1499-1510. doi: 10.1007/s00394-020-02343-9. Epub 2020 Jul 31. PMID 32737613
- [Background] Anderson JR, Hawkins MAW, Updegraff J, Gunstad J, Spitznagel MB. Baseline glucoregulatory function moderates the effect of dairy milk and fruit juice on postprandial cognition in healthy young adults. Eur J Nutr. 2018 Oct;57(7):2343-2352. doi: 10.1007/s00394-017-1505-0. Epub 2017 Jul 13. PMID 28707217
- [Background] Nabb SL, Benton D. The effect of the interaction between glucose tolerance and breakfasts varying in carbohydrate and fibre on mood and cognition. Nutr Neurosci. 2006 Jun-Aug;9(3-4):161-8. doi: 10.1080/10284150600955099. PMID 17176639
- [Background] Philippou E, Constantinou M. The influence of glycemic index on cognitive functioning: a systematic review of the evidence. Adv Nutr. 2014 Mar 1;5(2):119-30. doi: 10.3945/an.113.004960. PMID 24618754
- [Background] Smith MA, Riby LM, Eekelen JA, Foster JK. Glucose enhancement of human memory: a comprehensive research review of the glucose memory facilitation effect. Neurosci Biobehav Rev. 2011 Jan;35(3):770-83. doi: 10.1016/j.neubiorev.2010.09.008. Epub 2010 Sep 29. PMID 20883717
- [Background] Gaylor CM, Benton D, Brennan A, Young HA. The impact of glycaemic load on cognitive performance: A meta-analysis and guiding principles for future research. Neurosci Biobehav Rev. 2022 Oct;141:104824. doi: 10.1016/j.neubiorev.2022.104824. Epub 2022 Aug 11. PMID 35963545
- [Background] Benton D, Ruffin MP, Lassel T, Nabb S, Messaoudi M, Vinoy S, Desor D, Lang V. The delivery rate of dietary carbohydrates affects cognitive performance in both rats and humans. Psychopharmacology (Berl). 2003 Feb;166(1):86-90. doi: 10.1007/s00213-002-1334-5. Epub 2002 Dec 12. PMID 12488949
- [Background] Brand-Miller JC, Stockmann K, Atkinson F, Petocz P, Denyer G. Glycemic index, postprandial glycemia, and the shape of the curve in healthy subjects: analysis of a database of more than 1,000 foods. Am J Clin Nutr. 2009 Jan;89(1):97-105. doi: 10.3945/ajcn.2008.26354. Epub 2008 Dec 3. PMID 19056599
- [Background] Blaak EE, Antoine JM, Benton D, Bjorck I, Bozzetto L, Brouns F, Diamant M, Dye L, Hulshof T, Holst JJ, Lamport DJ, Laville M, Lawton CL, Meheust A, Nilson A, Normand S, Rivellese AA, Theis S, Torekov SS, Vinoy S. Impact of postprandial glycaemia on health and prevention of disease. Obes Rev. 2012 Oct;13(10):923-84. doi: 10.1111/j.1467-789X.2012.01011.x. Epub 2012 Jul 11. PMID 22780564
- [Background] Edefonti V, Rosato V, Parpinel M, Nebbia G, Fiorica L, Fossali E, Ferraroni M, Decarli A, Agostoni C. The effect of breakfast composition and energy contribution on cognitive and academic performance: a systematic review. Am J Clin Nutr. 2014 Aug;100(2):626-56. doi: 10.3945/ajcn.114.083683. Epub 2014 May 7. PMID 24808492
- [Background] Edefonti V, Bravi F, Ferraroni M. Breakfast and behavior in morning tasks: Facts or fads? J Affect Disord. 2017 Dec 15;224:16-26. doi: 10.1016/j.jad.2016.12.028. Epub 2016 Dec 24. PMID 28062077